CLINICAL TRIAL: NCT06868069
Title: Study on Blood Pressure Variability and Frailty in the Older People: the HypoPHrail Study
Brief Title: Study on Blood Pressure Variability and Frailty in the Older People
Acronym: HypoPHrail
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 09C409
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Old Age
Keywords: Blood pressure variability; Frailty
MeSH Terms: conditions — Hypertension; Frailty | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hypertension, aged 75 years and older
  Interventions: Diagnostic Test: Diagnostic tests and questionnaires

INTERVENTIONS:
Diagnostic Test: Diagnostic tests and questionnaires — Assessment of office blood pressure, orthostatic hypotension, 24-hour ambulatory blood pressure, frailty

SUMMARY:
Observational prospective single-center, non-profit study. Primary objective of the study: To determine if the hypotensive phenotype, defined as one episode of daytime systolic blood pressure (SBP) <90 mmHg (or two episodes of daytime SBP <90 mmHg, if mean 24 h SBP is <125 mmHg) detected at Ambulatory Blood Pressure Monitoring (ABPM) is associated with adverse events at follow up (death, hospitalization, falls, emergency room admission for uncontrolled hypertension, major cardiovascular events)

DETAILED DESCRIPTION:
Observational prospective single-center, non-profit study. Primary objective of the study: To determine if the hypotensive phenotype, defined as one episode of daytime systolic blood pressure (SBP) <90 mmHg (or two episodes of daytime SBP <90 mmHg, if mean 24 h SBP is <125 mmHg) detected at Ambulatory Blood Pressure Monitoring (ABPM) is associated with adverse events at follow up (death, hospitalization, falls, emergency room admission for uncontrolled hypertension, major cardiovascular events)

Secondary objectives of the study:

* To examine the association between home Blood Pressure Variability (BPV) and frailty, assessed using various tools for assessing frailty
* To examine the association between short term BPV and adverse events at follow up (death, hospitalization, falls, emergency room admission for uncontrolled hypertension, major cardiovascular events)
* To determine the prevalence of hypotensive phenotype according to frailty status in hypertensive individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Diagnosis of hypertension according to the criteria of the European Society of Cardiology guidelines [Williams 2018]
* Consent of the patient (or legal representative) to participate in the study

Exclusion Criteria:

* Refusal of the patient or his/her legal representative
* Life expectancy of less than 6 months

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly hypertensive patients who are enrolled at the Hypertension Centre of Istituto Auxologico italiano IRCCS
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | At 24 months of follow-up
  Adverse events at follow up (death, hospitalization, falls, emergency room admission for uncontrolled hypertension, major cardiovascular events)
Prevalence of hypotensive phenotype | At baseline
  Hypotensive phenotype, defined as one episode of daytime systolic blood pressure (SBP) <90 mmHg (or two episodes of daytime SBP <90 mmHg, if mean 24 h SBP is <125 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No